CLINICAL TRIAL: NCT01038726
Title: Neural Effects of Exercise, Cognitive, or Combined Training in AD At-Risk Elders
Brief Title: Effects of Exercise and Cognitive Training on Cognitive Function in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NIH AG035775-01
Record Dates: First submitted 2009-12-21; First posted 2009-12-24 (Estimated); Last update posted 2013-09-18 (Estimated); Status verified 2013-09

CONDITIONS: Aging; Alzheimer's Disease
Keywords: Healthy Aging
MeSH Terms: conditions — Alzheimer Disease | interventions — Exercise; Cognitive Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Exercise Training (Active Comparator)
  Interventions: Other: Exercise Training
- Combined Cognitive/Exercise Training (Active Comparator)
  Interventions: Other: Exercise Training; Other: Cognitive Training
- Cognitive Training (Active Comparator)
  Interventions: Other: Cognitive Training
- Combined Low Intensity Training (Active Comparator)
  Interventions: Other: Flexibility Training; Other: Educational Sessions

INTERVENTIONS:
Other: Exercise Training — Aerobic exercise training program designed by the Cardiac Rehabilitation department
  Arms: Combined Cognitive/Exercise Training; Exercise Training
Other: Cognitive Training — Based on cognitive training program Brain Fitness®
  Arms: Cognitive Training; Combined Cognitive/Exercise Training
Other: Flexibility Training — Non-aerobic flexibility training program designed by the Cardiac Rehabilitation department
  Arms: Combined Low Intensity Training
Other: Educational Sessions — DVD-based educational programs on history, art, and literature
  Arms: Combined Low Intensity Training

SUMMARY:
The purpose of this study is to gain a better understanding of the effects of exercise and cognitive training on improving brain function in healthy older adults who may be at risk for developing Alzheimer's Disease.

ELIGIBILITY:
Inclusion Criteria:

* First or Second-degree relative of someone with Alzheimer's Disease
* Not currently engaging in regular exercise
* Able to undergo an MRI
* Fluent in English

Exclusion Criteria:

* Neurological illnesses/conditions
* Medical illness/conditions that may affect brain function
* Any unstable or severe cardiovascular disease or asthmatic condition
* Severe depressive symptoms
* Inability to walk unassisted

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2009-12; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Brain activation patterns measured by functional MRI | baseline and 12 weeks

SECONDARY OUTCOMES:
Neuropsychological Testing | baseline and 12 weeks
Exercise assessment | baseline and 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Stephen M Rao, Ph.D., Principal Investigator — The Cleveland Clinic
Locations (1):
- The Cleveland Clinic, Cleveland, Ohio, United States